CLINICAL TRIAL: NCT02102412
Title: A Single-center Study to Evaluate the Safety & Performance of the Aer-O-Scope for Traveling Through the Colon in Healthy Volunteers
Brief Title: First in Man Aer-O-Scope
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Changes made to device.
Sponsor: GI View Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: 053 CLD ars 08
Record Dates: First submitted 2014-03-30; First posted 2014-04-02 (Estimated); Last update posted 2017-08-01 (Actual); Status verified 2014-03

CONDITIONS: Screening Colonoscopy for Low Risk Subjects
Keywords: crc; colonoscopy; colon cancer
MeSH Terms: conditions — Colonic Neoplasms | interventions — Colonoscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- single arm (Experimental): single arm patients underwent colonoscopy with aer-o-scope followed by conventional colonoscopy to assess if any mucosal damage occurred with the experimental device.
  Interventions: Biological: screening colonoscopy

INTERVENTIONS:
Biological: screening colonoscopy — performance of a colonoscopy with the experimental device followed by complete conventional colonoscopy
  Other Names: colonoscopy

SUMMARY:
A single center study intended to evaluate the Aer-O-Scope Colonoscope System.

DETAILED DESCRIPTION:
A clinical study in Zagreb Croatia, intended to evaluate the Aer-O-Scope Colonoscope System. The study includes 120 subjects and has the following endpoints:

Evaluation of the Aer-O-Scope advancement, imaging and retraction throughout the Colon.

Safety: No occurrence of any device related major adverse event (for details see section 9.5)

Efficacy:

1. Advancement of device towards the ceacum and retraction
2. Visualization of the colon mucosa by the traveling imaging device
3. Procedure duration
4. Handling and operation (assessment by operator)

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers between 18 and 65 years of age.
* Sign informed consent.

Exclusion Criteria:

* Subjects with any known GI related symptoms complaints or GI diseases.
* Subjects with cancer or other life threatening diseases or conditions.
* Pregnant women.
* Subjects who underwent any abdominal surgery.
* Morbid Obesity (BMI > 40).
* Drug abuse or alcoholism.
* Bed-ridden subject.
* Inadequate communication with the subject.
* Subjects under custodial care.
* Participation in any clinical study within the last 30 days.
* Subjects with known cardiovascular and pulmonary diseases.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 101 (Actual)
Dates: Start 2005-02; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
Ability to traverse the colon using the aer-o-scope | under 60 minutes
  a propulsion system using low pressure co2 gas and balloons is used to propel the system through the colon

CONTACTS AND LOCATIONS:
Overall Officials: Boris Vucelic, MD, Principal Investigator — Chief Gastro, Zagreb
Locations (1):
- Rebro Hospital, Zagreb, Croatia